CLINICAL TRIAL: NCT04767880
Title: Acute Metabolic Effects of Pre-meal Consumption of Whey in Women at Risk of Gestational Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 1-10-72-305-20
Record Dates: First submitted 2021-02-12; First posted 2021-02-23 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2022-05

CONDITIONS: Gestational Diabetes Mellitus in Pregnancy
MeSH Terms: interventions — Whey

STUDY DESIGN:
Intervention Model Description: Singleblind, randomized, crossover design
Who Masked: Participant
Masking Description: Participants will be blinded to the intervention and placebo in the laboratory setting.
  Quadruple (Participants, care providers, investigators and outcome assessors) Participants, care providers, investigators and outcome assessors will be blinded to the placebo and varying doses of whey in the home setting.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Whey (Experimental): Whey protein isolate WPI (Lacprodan® ISO.Water. from Arla Foods Ingredients). The intervention will be ingested 30 min. prior to an OGTT (3 hours). The intervention will also be ingested 30 min prior to breakfast in the women's own environment.
  Interventions: Dietary Supplement: Whey
- Placebo (Placebo Comparator): The placebo will be ingested 30 min. prior to an OGTT (3 hours). The placebo will also be ingested 30 min prior to breakfast in the women's own environment.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Whey — Doses of 10, 15, 20 and 30 gram protein of a regular whey protein compound (whey protein isolate WPI (Lacprodan® ISO.Water. from Arla Foods Ingredients))
  Arms: Whey
Dietary Supplement: Placebo — The placebo contains <1 kcal and 0 g protein
  Arms: Placebo

SUMMARY:
The main objective of our study is to investigate the metabolic effects of whey protein (whey protein isolate, WPI, (Lacprodan® ISO.Water. from Arla Foods Ingredients) compared to placebo when consumed by women in risk of gestational diabetes mellitus (GMD) 30 minutes prior to an oral glucose tolerance test (OGTT). We will also investigate any changes in substrate metabolism and energy expenditure using indirect calorimetry. Differences in hunger and satiety parameters as well as rate of gastric emptying will also be assessed. Furthermore, we will investigate the glucose response when the women consume the intervention at home in their own environment 30 minutes before breakfast in various doses (placebo, 10, 15, 20, 30 g whey). The women will be monitored with continuous glucose monitors, activity monitors and all meals will be provided.

The two study days in the laboratory will be repeated 3-9 months after pregnancy. The purpose of this is to be able to compare the metabolic response of pre-meal whey during pregnancy with the response in a not-pregnant state. The study days at home will not be repeated after pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Referred to screening for Gestational Diabetes Mellitus by week 24-30 or GDM
* BMI 20-35
* Normal blood pressure
* Age > 18 years

Exclusion Criteria:

* Special dietary regimes > 1 month at time of inclusion e.g. ketogenic diet
* Daily intake of protein supplements
* Milk allergy or phenylketonuria
* Celiac disease
* Medication with effect on glucose metabolism e.g. steroid
* Do not speak or understand Danish
* Gemelli
* Polycystic Ovarian Syndrome
* PI finds the patient unfit (like mental illness, too nervous or other)
* Anemia (hemoglobin <6 mmol/l)
* Severe chronic illness
* Depression
* Severe nausea/vomiting
* Non-breakfast eaters

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-04-26 (Actual); Primary Completion 2023-09-29 (Actual); Study Completion 2023-09-29 (Actual)

PRIMARY OUTCOMES:
Concentration differences in blood glucose following an OGTT | 3 hours following the OGTT

SECONDARY OUTCOMES:
Concentration differences in glucose independent peptide (GIP) | 3 hours following the OGTT
Concentration differences in glucagon like peptide 1 (GLP-1) | 3 hours following the OGTT
Concentration differences in glucagon | 3 hours following the OGTT
Concentration differences in insulin | 3 hours following the OGTT
Concentration differences in c-peptide | 3 hours following the OGTT
Concentration differences in free fatty acids (FFA) | 3 hours following the OGTT
Concentration differences in ghrelin | 3 hours following the OGTT
Concentration differences in leptin | 3 hours following the OGTT
Concentration differences in amino acids (AA) | 3 hours following the OGTT
Gastric emptying rate (Concentration differences in blood paracetamol/acetaminophen) | 3 hours following the OGTT
Resting energy expenditure (REE) (Resting Metabolic Rate) | 3 hours following the OGTT
Respiratory quotient (RQ) | 3 hours following the OGTT
Self-reported appetite | 3 hours following the OGTT and 3 hours following breakfast
  A visual analogue scale ranging from "not at all" to "extremely" will be used to assess Hunger, Fullness, Satiety, Desire, Prospective consumption (Quantity).
Heart rate | 5 days
  A combined accelerometer and heart rate monitor will be used to measure heart rate (beats/minute)
Energy expenditure | 5 days
  A combined accelerometer and heart rate monitor will be used to estimate energy expenditure (kCal)
Activity | 5 days
  A combined accelerometer and heart rate monitor will be used to measure activity (counts/minute)
Continuous glucose measurements (CGM) | 5 days
  Time in range, concentration differences in interstitial fluid glucose 3 hours following breakfast, glycemic variability, mean glucose, daily maximum glucose, estimated HbA1c

CONTACTS AND LOCATIONS:
Overall Officials: Per G Ovesen, Professor, Study Director — Institute of Clinical Medicine, Aarhus University and Department of Gynecology and Obstetrics and Steno Diabetes Center Aarhus, Aarhus University Hospital
Locations (1):
- Medicinsk forskningslaboratorium for Diabetes og Hormonsygdomme og Steno Diabetes Center Aarhus (M-lab), Aarhus universitetshospital, Aarhus, Denmark

REFERENCES:
- [Derived] Smedegaard S, Rittig N, Ovesen PG, Suder LB, Knudsen JH, Brunsgaard LH, Kampmann U. Once-daily supplementation with pre-meal whey protein lowers breakfast postprandial glucose levels in women with GDM throughout the third trimester: a randomised, controlled, clinical trial. Diabetologia. 2026 Feb;69(2):350-363. doi: 10.1007/s00125-025-06587-0. Epub 2025 Nov 7. PMID 41203981